CLINICAL TRIAL: NCT04131920
Title: Handheld Ultrasound (HHUS) for Home Use in Hemophilia
Acronym: HHUS
Status: Completed | Type: Observational
Sponsor: Washington Institute for Coagulation (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Kruse-Jarres, MD, MPH, Executive/Medical Director, Washington Center for Bleeding Disorders, Washington Institute for Coagulation
Other Study IDs: ML41066
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Joint Bleed; Hemophilia A
Keywords: Joint Bleed; Hemophilia A; Handheld Ultrasound
MeSH Terms: conditions — Hemarthrosis; Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Phase 1 and 2: 10 male patients with severe Hemophilia A from the Washington Center for Bleeding Disorders
  Interventions: Device: handheld ultrasound: Philips Lumify integrated tele-ultrasound powered by Reacts collaborative platform
- Phase 3: 20 subjects who are also participating in the EmiMSKUS study
  Interventions: Device: handheld ultrasound: Philips Lumify integrated tele-ultrasound powered by Reacts collaborative platform

INTERVENTIONS:
Device: handheld ultrasound: Philips Lumify integrated tele-ultrasound powered by Reacts collaborative platform — Patients receive training by the physical therapist to operate a handheld ultrasound (HHUS) including proper probe placement. Subjects will be tested on their knowledge at the HTC to demonstrate proficiency, and will then repeat the testing at home via tele-ultrasound.

SUMMARY:
This is a study in 3 phases that will assess the feasibility and utility of handheld home ultrasound (HHUS) in a patient's home to assess whether a painful episode in the elbow, knee or ankle is a bleed or not.

DETAILED DESCRIPTION:
This is a study in 3 phases that will assess the feasibility and utility of handheld home ultrasound (HHUS) in a patient's home to assess whether a painful episode in the elbow, knee or ankle is a bleed or not.

Phase 1 will assess whether 10 subjects with severe hemophilia A can be trained to use HHUS in clinic to identify basic joint structures of the elbow, knee and ankle. It will then assess whether these subjects can identify these structures at home and transmit the images life via tele-ultrasound.

Phase 2 will assess whether the determination of "bleed" vs. "non-bleed" made at home via HHUS can be confirmed/validated with a standard high resolution ultrasound machine in clinic.

Phase 3 will then utilize HHUS during the EmiMSKUS study over 3 years to more objectively identify patient reported bleeding during the study.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A
* Male
* Over 18 years of age
* Able to read, write and understand English
* Willing to come to the center for an 8 hour training session
* Lives in proximity of the HTC and is willing to come in for acute joint episodes in phase 2
* Willing and able to follow study procedures
* Willing and able to keep HHUS at a safe place
* Have the dexterity to operate a HHUS unit

Exclusion Criteria:

* Unable to follow study instructions
* Physically or mentally unable to operate a HHUS unit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males patients at Hemophilia Treatment Centers with severe Hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Outcome 1.1: Participant understanding of basic ultrasound transducer concepts and ability to perform basic positioning maneuvers. | 3 months
  Number of participating subjects who understand basic ultrasound transducer concepts and can perform basic positioning maneuvers based on post-training test.
Outcome 1.2: Participating subjects are able to perform basic transducer positions and identify basic structures of the elbow, knee and ankle. | 3 months
  Number of participating subjects who are able to perform basic transducer positions and identify basic structures of the elbow, knee and ankle based on post-training test.
Outcome 1.3: Participating subjects can perform what they learned during their training at the HTC in outcome 1.1 and outcome 1.2 at home and transmit images to the HTC. | 3 months
  Number of participating subjects who can perform what they learned during their training at the HTC in outcome 1.1 and outcome 1.2 at home and transmit images to the HTC on post-training test.
Outcome 2.1: Subjects will be able to attain and transmit images of their joint spaces to the HTC via telemedicine utilizing the HHUS technology they learned in phase 1 and React App. | 6 months
  Number of subjects who will be able to attain and transmit images of their joint spaces to the HTC via telemedicine utilizing the HHUS technology they learned in phase 1 and React App.
Outcome 2.2: Accuracy of the assignment of "bleed" vs. "non-bleed" will be determined on the stationary GE LS8 Logiq Pro in the HTC. | 6 months
  Percentage accuracy of the assignment of "bleed" vs. "non-bleed" will be determined on the stationary GE LS8 Logiq Pro in the HTC.
Outcome 3.1: To establish how accurate patient reported bleeding is compared to HHUS utilizing tele-ultrasound. | 3 years
  Percentage accuracy of patient reported bleeding is compared to HHUS utilizing tele-ultrasound.
Outcome 3.2: To establish more accurate bleeding data for the EmiMSKUS study. | 3 years
  Number of patients who have joint bleeding data incorporated into the EmiMSKUS study.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kruse-Jarres, MD, MPH, Principal Investigator — Washington Institute for Coagulation
Locations (1):
- Washington Center for Bleeding Disorders at Washington Institute for Coagulation, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forsyth AL, Giangrande P, Hay CR, Kenet G, Kessler CM, Knobl PN, Llinas A, Santagostino E, Young G. Difficult clinical challenges in haemophilia: international experiential perspectives. Haemophilia. 2012 Jul;18 Suppl 5:39-45. doi: 10.1111/j.1365-2516.2012.02887.x. PMID 22757683
- [Background] Manco-Johnson MJ, Abshire TC, Shapiro AD, Riske B, Hacker MR, Kilcoyne R, Ingram JD, Manco-Johnson ML, Funk S, Jacobson L, Valentino LA, Hoots WK, Buchanan GR, DiMichele D, Recht M, Brown D, Leissinger C, Bleak S, Cohen A, Mathew P, Matsunaga A, Medeiros D, Nugent D, Thomas GA, Thompson AA, McRedmond K, Soucie JM, Austin H, Evatt BL. Prophylaxis versus episodic treatment to prevent joint disease in boys with severe hemophilia. N Engl J Med. 2007 Aug 9;357(6):535-44. doi: 10.1056/NEJMoa067659. PMID 17687129
- [Background] Konkle BA, Ebbesen LS, Erhardtsen E, Bianco RP, Lissitchkov T, Rusen L, Serban MA. Randomized, prospective clinical trial of recombinant factor VIIa for secondary prophylaxis in hemophilia patients with inhibitors. J Thromb Haemost. 2007 Sep;5(9):1904-13. doi: 10.1111/j.1538-7836.2007.02663.x. PMID 17723130
- [Background] Leissinger C, Gringeri A, Antmen B, Berntorp E, Biasoli C, Carpenter S, Cortesi P, Jo H, Kavakli K, Lassila R, Morfini M, Negrier C, Rocino A, Schramm W, Serban M, Uscatescu MV, Windyga J, Zulfikar B, Mantovani L. Anti-inhibitor coagulant complex prophylaxis in hemophilia with inhibitors. N Engl J Med. 2011 Nov 3;365(18):1684-92. doi: 10.1056/NEJMoa1104435. PMID 22047559
- [Background] Oldenburg J, Mahlangu JN, Kim B, Schmitt C, Callaghan MU, Young G, Santagostino E, Kruse-Jarres R, Negrier C, Kessler C, Valente N, Asikanius E, Levy GG, Windyga J, Shima M. Emicizumab Prophylaxis in Hemophilia A with Inhibitors. N Engl J Med. 2017 Aug 31;377(9):809-818. doi: 10.1056/NEJMoa1703068. Epub 2017 Jul 10. PMID 28691557
- [Background] Mahlangu et al. Emicizumab prophylaxis administered once-weekly or every two weeks provides effective bleed prevention in persons with haemophilia A without inhibitors - Results from the phase III HAVEN 3 study . Oral presented at the World Federation of Hemophilia Meeting in Glasgow, May 21, 2018.
- [Background] Ceponis A, Wong-Sefidan I, Glass CS, von Drygalski A. Rapid musculoskeletal ultrasound for painful episodes in adult haemophilia patients. Haemophilia. 2013 Sep;19(5):790-8. doi: 10.1111/hae.12175. Epub 2013 May 15. PMID 23672827
- [Background] Zhou JY, Rappazzo KC, Volland L, Barnes RFW, Brackman M, Steiner B, Kruse-Jarres R, Quon DV, Bailey C, Chang EY, von Drygalski A. Pocket handheld ultrasound for evaluation of the bleeding haemophilic joint: A novel and reliable way to recognize joint effusions. Haemophilia. 2018 Mar;24(2):e77-e80. doi: 10.1111/hae.13429. Epub 2018 Feb 12. No abstract available. PMID 29436079